CLINICAL TRIAL: NCT00319839
Title: A Phase II Study of Albumin Bound-Paclitaxel (AbraxaneTM) for Treatment of Recurrent or Metastatic Head and Neck Cancer With the Addition of Cetuximab (Erbitux) (IMC-225) on Disease Progression
Brief Title: Study of Albumin Bound-Paclitaxel for Treatment of Recurrent or Metastatic Head and Neck Cancer With Cetuximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sai-Hong Ignatius Ou, HS Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 05-46; 2005-4667 (Other: University of California, Irvine)
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Cancer
Keywords: Head cancer; Neck cancer; cetuximab; abraxane; erbitux; IMC-225; NSC-714692
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Albumin-Bound Paclitaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane plus Cetuximab (Experimental): Drug: Abraxane-260 mg/m2 IV over 30 minutes every 3 weeks. Drug: Cetuximab will be added to Abraxane if there is documented progression on single agent Abraxane. First dose: 400 mg/m2 IV over 120 minutes. Weekly: 250 mg/m2 IV over 60 minutes Days 8 and 15 of cycle 1 and days 1, 8, 15 of all subsequent cycles.
  Interventions: Drug: Abraxane; Drug: Cetuximab

INTERVENTIONS:
Drug: Abraxane — 260 mg/m2 IV over 30 minutes every 3 weeks
  Other Names: Albumin-bound Paclitaxel; ABI-007
Drug: Cetuximab — Cetuximab will be added to Abraxane if there is documented progression on single agent Abraxane. First dose: 400 mg/m2 IV over 120 minutes. Weekly: 250 mg/m2 IV over 60 minutes Days 8 and 15 of cycle 1 and days 1, 8, 15 of all subsequent cycles
  Other Names: IMC-225; Erbitux; NSC-714692

SUMMARY:
Primary Objective: To assess the overall response rate (complete and partial response) to Abraxane in patients with recurrent or metastatic head and neck cancer with the addition of Cetuximab on disease progression.

Approximately 40,000 new cases of head and neck cancer are diagnosed annually in the United States (Jemal et al, 2003), and over 30% of these patients are expected to die of their malignancy. Squamous cell carcinoma accounts for more than 90% of head and neck cancer cases. Although metastatic disease at the time of diagnosis is rather uncommon, and despite aggressive use of up-front concurrent radiation and cisplatin-based chemotherapy, approximately 20% of the patients will develop metastases. Patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) have a poor prognosis

A subsequent randomized study conducted by ECOG (E1393) compared high-dose paclitaxel (200 mg/m2) as a 24-hour infusion plus cisplatin 75 mg/m2 with G-CSF support, to low dose paclitaxel (135 mg/m2) as a 24-hour infusion, plus cisplatin 75 mg/m2 (Forastiere et al, 2001). Patients with newly diagnosed metastatic or recurrent squamous cell carcinoma of the head and neck, excluding nasopharyngeal primaries were eligible. No prior treatment for recurrent/metastatic disease was allowed, but patients could have received chemotherapy as a part of the initial curative therapy that should have been completed 6 months prior to study.

No statistically significant difference could be demonstrated either in response rates or survival between the two arms (Murphy et al, 2001). This study, however, indicated that paclitaxel, a member of the taxane class of anti-tumor agent, is active in head and neck cancer.

New agents to treat head and neck cancer need to be investigated. Abraxane, an albumin-bound formulation of paclitaxel has shown significant single-agent activity in breast cancer and in head and neck cancer. Recently, Abraxane has approved for use in metastatic breast cancer. Given previous randomized phase III trials indicated single agent chemotherapy fared as well as combination chemotherapy regimen in terms of overall survival, this novel formulation should be actively investigated in head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objective: To assess the overall response rate (complete and partial response) to Abraxane in patients with recurrent or metastatic head and neck cancer with the addition of Cetuximab on disease progression.

Secondary Objectives: 1. To assess the frequency and severity of toxicities associated with this treatment. 2. To evaluate overall survival and progression-free survival in patients with recurrent or metastatic head and neck cancer treated with single agent Abraxane. 3.To assess whether the addition of Cetuximab will re-sensitize head and neck cancer to Abraxane after progression on single agent Abraxane.

BACKGROUND AND RATIONALE

Approximately 40,000 new cases of head and neck cancer are diagnosed annually in the United States (Jemal et al, 2003), and over 30% of these patients are expected to die of their malignancy. Squamous cell carcinoma accounts for more than 90% of head and neck cancer cases. Although metastatic disease at the time of diagnosis is rather uncommon, and despite aggressive use of up-front concurrent radiation and cisplatin-based chemotherapy, approximately 20% of the patients will develop metastases. Patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) have a poor prognosis. Their median survival is about 6-8 months. Selected patients with locally recurrent disease can be treated with a curative intent with locoregional therapies, such as salvage surgery or radiation (De Crevoisier et al, 1998); however the majority of these patients die of their disease. Despite high response rates, combination chemotherapy has not been shown to produce a survival benefit compared to single agents in randomized trials in patients with recurrent/metastatic head and neck cancer (Forastiere et al, 1992; Jacobs et al, 1992; Clavel et al, 1994). A phase III randomized study conducted by Southwest Oncology Group (SWOG) compared cisplatin-based combination chemotherapy to single agent methotrexate (Forastiere et al, 1992). The objective response rates were 32%, 21%, and 10%, for cisplatin/5-Fluorouracil (5-FU), carboplatin/5-FU, and single methotrexate, respectively, but the median overall survival was not statistically different between the three arms (ranged between 5 to 6.6 months). Moreover, toxicity was increased with combination therapy, especially with the cisplatin-based regimen. Another randomized study conducted in the US demonstrated a significantly higher response rate of 32% for the combination of cisplatin and 5-FU versus 17% and 13% for single agent cisplatin and 5-FU, respectively (Jacobs et al, 1992). However, the median survival of all patients was 5.7 months, with no difference between the three arms. Hematologic toxicity was increased in the combination arm.

A subsequent randomized study conducted by ECOG (E1393) compared high-dose paclitaxel (200 mg/m2) as a 24-hour infusion plus cisplatin 75 mg/m2 with granulocyte-colony stimulating factor (G-CSF) support, to low dose paclitaxel (135 mg/m2) as a 24-hour infusion, plus cisplatin 75 mg/m2 (Forastiere et al, 2001). Patients with newly diagnosed metastatic or recurrent squamous cell carcinoma of the head and neck, excluding nasopharyngeal primaries were eligible. No prior treatment for recurrent/metastatic disease was allowed, but patients could have received chemotherapy as a part of the initial curative therapy that should have been completed 6 months prior to study. Tow hundred and ten patients were randomized between the 2 arms. No significant difference in outcome was observed. The response rate was 35% vs 36% and the median survival was 7.6 vs 6.8 months, in the high-dose vs low-dose paclitaxel arms respectively. Patients with metastatic disease performed worse in terms of survival. Previously untreated patients achieved a higher response rate of 58% compared to a response rate of 32% observed in patients who have failed prior curative therapies. Substantial toxicities were observed in this trial. Grade 4 neutropenia was seen in 61-71% of patients and febrile neutropenia with hospitalization occurred in 27-39% of patients. The toxic death rate was 10% (12% vs 9%) (Forastiere et al, 2001). It was concluded that the 24-hour paclitaxel infusion was associated with unacceptable toxicity when combined with cisplatin. Instead, a 3-hour paclitaxel infusion combined with cisplatin was advanced to further testing. A more recent randomized trial conducted by ECOG (E1395) compared the combination of paclitaxel 175 mg/m2 as a 3-hour infusion and cisplatin 75 mg/m2 to a standard cisplatin and 5-FU regimen. No statistically significant difference could be demonstrated either in response rates or survival between the two arms (Murphy et al, 2001). This study, however, indicated that paclitaxel, a member of the taxane class of anti-tumor agent, is active in head and neck cancer.

Recently, another member anti-tumor class of taxane, Docetaxel (Taxotere) has been shown to be active in advanced head and neck cancer. In a randomized phase III trial of intensification of induction chemotherapy followed by radiation, the addition of docetaxel to the induction regimen of cisplatin and 5-fluoruracil when compared to cisplatin and 5-fluoruracil alone resulted in a 3-month improvement in overall survival (Vermorken et al, 2004). Thus both members of the taxane family, paclitaxel and docetaxel, have proven anti-tumor activity in head and neck cancer.

New agents to treat head and neck cancer need to be investigated. Abraxane, an albumin-bound formulation of paclitaxel has shown significant single-agent activity in breast cancer and in head and neck cancer. Recently, Abraxane has approved for use in metastatic breast cancer. Given previous randomized phase III trials indicated single agent chemotherapy fared as well as combination chemotherapy regimen in terms of overall survival, this novel formulation should be actively investigated in head and neck cancer.

Abraxane in solid tumor The clinical database included two single arm studies enrolling a total of 106 patients and one multi-center randomized trial. The multi-center trial was conducted in 460 patients with metastatic breast cancer who were randomized to receive either Abraxane 260 mg/m² administered as a 30-minute infusion or paclitaxel 175 mg/m² given over 3 hours. Sixty-four percent of patients had impaired performance status (ECOG 1 or 2) at study entry. Seventy-nine percent had visceral metastases and 76% had > 3 sites of metastases. Fifty-nine percent of patients had received one or more prior chemotherapy regimens, and 77% had received an anthracycline-containing regimen. The objective response rate verified by central review was 21.5% (95% Confidence interval (CI): 16.2% to 26.7%) for Abraxane compared to 11.1% (95% CI: 6.9% to 15.1%) for paclitaxel (p=0.003). The conclusion of this phase III trial is that Abraxane had statistically significant higher target lesion response rate (the trial primary endpoint) (O'Shaughnessy et al, 2003).

On January 7, 2005 the U. S. Food and Drug Administration approved Abraxane (albumin-bound paclitaxel) for treatment of breast cancer after failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy based on the statistically significant superior response rate from the randomized phase III trial mentioned above. The recommended dose of Abraxane is 260 mg/m² administered intravenously over 30 minutes every 3 weeks. No premedication to prevent hypersensitivity reactions is required prior to Abraxane administration.

Abraxane in Head and Neck Cancer The role of Abraxane in Head and Neck cancer has been explored in a phase I study (Damascelli et al, 2001). Abraxane was injected intra-arterially (carotid artery) in 31 patients with advanced Head and Neck cancer. The maximum tolerated dose in a single administration was determined to be 270 mg/m2 which is very close to the approved dose of 260 mg/m2. Three patients achieved complete response and 19 patients achieved partial response for a combined response rate of 76%. Side effects are very tolerable including three patients with grade 4 neutropenia, and grade 2 non-hematologic toxicities included: keratitis [1 patient], skin toxicity [5 patients], neurologic toxicities [4 patients], and flu-like syndrome [7 patients]. However, intra-arterial administration is technically challenging with potential serious side effects, cumbersome and not the conventional way of delivering chemotherapy. In another phase 1 study of Abraxane in advanced solid tumors, 3 out of 5 patients with nasopharyngeal carcinoma had responses lasting 25, 18 and 13+ weeks (Teng et al, 2005).

Given the hint of anti-tumor activity of Abraxane in advanced Head and Neck cancer from the above mentioned studies, this current study will seek to determine the efficacy of Abraxane in recurrent or metastatic head and neck cancer at the dose of 260 mg/m2 given intravenously every 3 weeks in a systemic manner. Abraxane is not FDA approved in the treatment of this study disease; however, it is approved for patient use in the treatment of advanced breast cancer that have failed traditional therapy.

Abraxane is a natural substance and is far more superior to conventional chemistry. Abraxane is an effective treatment for aggressive cancers because it adversely affects the process of cell division by preventing this restructuring. Other cells are also affected adversely, but since cancer cells divide much faster than non-cancerous cells, they are far more susceptible to Abraxane treatment, thus, the safety of the drug is no more or less then other chemotherapy regimens.

Human albumin will be used along with the Abraxane.

Description of Cetuximab (IMC-225) (Erbitux) (NSC-714692) Cetuximab, a chimerized antibody of the immunoglobulin gamma-1 (IgG1) subclass was originally derived from a mouse myeloma cell line. The chimerization resulted in an antibody with binding affinity to epidermal growth factor receptors (EGFR) greater than the natural ligand epidermal growth factor (EGF). Cetuximab blocks binding EGF and transforming growth factor (TGFa) to EGFR and inhibits ligand-induced activation of this tyrosine kinase receptor. Cetuximab also stimulates EGFR internalization, effectively removing the receptor from the cell surface for interaction with ligand.

Safety Precaution Cetuximab therapy should be used with caution in patients with known hypersensitivity to Cetuximab, murine proteins, or any component of this product.

Administration of Cetuximab: In an effort to prevent a hypersensitivity reaction, all patients should be premedicated with dexamethasone 20 mg by IV and diphenhydramine hydrochloride 50 mg by IV given 30-60 minutes prior to the infusion of cetuximab.

The initial/loading dose of cetuximab is 400 mg/m2 IV administered over 120 minutes. Patients must be continuously observed during the infusion for signs of anaphylaxis and standard resuscitative meds should be in close proximity. Vital signs should be taken prior to, during, post and 1-hour post infusion for the initial dose. For subsequent infusions, vital signs are recommended to be taken to and 1-hour post infusion.

Following the loading dose, patients will receive weekly treatment with cetuximab IV over 60 minutes. The infusion rate of cetuximab should never exceed 5 mL/min. Patients should be closely monitored for treatment-related adverse events, especially hypersensitivity reactions, during the infusion and post-infusion.

Cetuximab is used for the treatment of patients with advanced head and neck cancer that has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed carcinoma of the head and neck region. Primary tumor sites include: lip and oral cavity, major salivary glands, pharynx (oropharynx, nasopharynx, hypopharynx), or larynx (supraglottis, glottis, subglottis), nasal cavity and paranasal sinuses, and thyroid
* Patients must have metastatic or locally recurrent squamous cell carcinoma of the head and neck. Patients with locoregional disease must be considered incurable by means of locoregional therapy.
* All sites of disease must be assessed and designated as measurable or non-measurable disease as documented by CT, MRI, X-ray physical exam or nuclear exam. All measurable and non-measurable disease must be assessed within 28 days prior to registration.
* Patients may have prior chemotherapy for recurrent/metastatic disease. However, all chemotherapy must be completed at least 21 days prior to scheduled start of Abraxane.
* Patients must have adequate bone marrow reserve as documented by absolute neutrophil count (ANC) > 1,500 μl and platelets > 100,000/ μl obtained within 14 days prior to registration.
* Patients must have adequate hepatic as documented by serum bilirubin < 1.5 x the institutional upper limit of normal. These tests must be obtained within 14 days prior to registration.
* All patients must be 18 years of age or older
* Patients must have a Zubrod performance of 0-3

Exclusion Criteria:

* Patients must not have prior therapy with Abraxane
* Patients with any evidence of active or uncontrolled infection, recent myocardial infection, unstable angina, or life-threatening arrhythmia are not eligible.
* Patients with baseline grade 3 peripheral neuropathy are not eligible.
* Patients with known brain metastasis are not eligible. However, brain-imaging studies are not required for eligibility if the patient has no neurological signs or symptoms. If brain-imaging studies are performed, they must be negative for disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S.-H. Ignatius Ou, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: March 2006 Primary completion date: May 2009 Study completion date: June 2010
Period: Overall Study
Arm/Group | Abraxane Plus Cetuximab
Started | 7
Completed | 1
Not Completed | 6
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane Plus Cetuximab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Response)
Description: To assess the overall response rate (complete and partial response) to Abraxane in patients with recurrent or metastatic head and neck cancer.
Time Frame: 3 years
Population: Analysis was not completed as the study was terminated early due to low accrual and of the 7 subjects who went on study, only 1 completed treatment.
Arm/Group | Abraxane Plus Cetuximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency and Severity of Toxicities
Description: To assess the frequency and severity of toxicities associated with this treatment.
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Abraxane Plus Cetuximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival and Progression-free Survival in Patients
Time Frame: 3 years
Arm/Group | Abraxane Plus Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years, 1 month
Arm/Group | Abraxane Plus Cetuximab
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane Plus Cetuximab (N=7)
Influenza Grade III (General disorders) | 1 — Hospital admission for fever, chills, cough with sputum, and WBC count of 1,000/mcl.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane Plus Cetuximab (N=7)
Constipatoin (Gastrointestinal disorders) | 1
Difficulty Breathing and Swallowing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes